CLINICAL TRIAL: NCT01127880
Title: The Role of Antibiotics in the Reduction of Infectious Complications in Tube Thoracotomy Management of Traumatic Hemopneumothorax: A Prospective, Double-Blinded Study
Brief Title: Role of Antibiotics to Reduce Infectious Complications in Tube Thoracotomy Management of Traumatic Hemopneumothorax
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Nathaniel McQuay, Jr., MD, St. Luke's Hospital and Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SLHN 2005-34
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2009-02

CONDITIONS: Hemopneumothorax; Pneumothorax
Keywords: Traumatic Hemopneumothorax; Thoracotomy; Antibiotics
MeSH Terms: conditions — Hemopneumothorax; Pneumothorax | interventions — Cefazolin; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ancef 1 gm or Clindamycin 300 mg (Active Comparator): Group A will receive Ancef 1gm or Clindamycin 300mg if penicillin or bet-lactam allergy exists
  Interventions: Drug: Ancef or Clindamycin
- Placebo (Placebo Comparator): Group B will receive .9% Normal Saline as a placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ancef or Clindamycin — 1 gm of Ancef or 300 mg Clindamycin for those who are penicillin allergic
  Arms: Ancef 1 gm or Clindamycin 300 mg
Drug: Placebo — .9% Normal Saline as a placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the efficacy of prophylactic antibiotics in patients with chest tubes for management of thoracic injuries in the reduction of the incidence of empyema as compared to placebo.

DETAILED DESCRIPTION:
In this study, the medication (an antibiotic which is used to treat or prevent infections) will be compared with a placebo. A placebo is something that looks like a "real" medication, but it doesn't contain any active medication. As a participant in this study, you may receive the active medication (Cefazolin Sodium Injection or Clindamycin) or you may receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years of age.
2. Admission to Trauma, General Surgery, and/or Surgical Critical Care services.
3. Traumatic pneumothorax, hemothorax or hemopneumothorax

Exclusion Criteria:

1. Pregnancy
2. Open fracture
3. Immunocompromised
4. Require antibiotics for treatment of other injuries
5. Chest tube placement greater than 72hrs after admission

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
efficacy of prophylactic antibiotics in reduction of empyema | 30 days
  The primary objective of this study is to examine the efficacy of prophylactic antibiotics in patients with chest tubes for management of thoracic injuries in the reduction of the incidence of empyema as compared to placebo.

SECONDARY OUTCOMES:
Incidence of Pneumonia and/or development of resistant microorganisms | 30 days
  Secondary objectives include:
  Incidence of pneumonia Incidence of development of resistant microorganisms

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel McQuay, MD, Principal Investigator — St. Luke's Hospital and Health Network
Locations (1):
- St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania, United States